CLINICAL TRIAL: NCT03390933
Title: Using Latent Variables and Directly Observed Treatment to Improve the Diagnosis and Management of Depression Among Hemodialysis Patients
Brief Title: Identifying and Treating Depression in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Ash Sehgal, Principal Investigator, MetroHealth Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-00768
Record Dates: First submitted 2017-10-12; First posted 2018-01-05 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Depression; Hemodialysis-Induced Symptom
MeSH Terms: conditions — Depression | interventions — Fluoxetine

STUDY DESIGN:
Intervention Model Description: The cross-sectional study will involve assessments of depressive symptoms (PHQ-9) and quality of life for 1083 patients. These data will be used to address Aim A. The single arm trial will involve 96 patients with DSM5-confirmed depression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fluoxetine Group (Experimental): Approximately 96 patients will be enrolled into the intervention (Phase II) over the duration of the entire study.
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine — Patients enrolled into Phase II will be prescribed 2 weeks of short-acting fluoxetine 20 mg and will be instructed to take the prescription daily for 2 weeks. Then patients will be prescribed 10 additional weeks of 90 mg (weekly) fluoxetine and will be observed taking it once weekly at the dialysis unit. At the end of the 12 week study period, participants will be provided 4 additional weeks of 90 mg fluoxetine in order to provide sufficient time to follow up with their primary care physician or nephrologist.
  Other Names: Prozac

SUMMARY:
Depression is present in about 20-30% of hemodialysis patients and is associated with morbidity and mortality. However, depression is inadequately diagnosed and treated among dialysis patients. This is due in part to the overlap between depressive symptoms (e.g. appetite change, trouble sleeping, feeling tired) and symptoms related to persistent metabolic derangements in hemodialysis patients (e.g. nausea, nocturnal cramps, feeling washed out after treatment). The overlap between depressive symptoms and dialysis-related complications makes it difficult to diagnose and therefore to treat depression. In addition, prescription of antidepressant medication may increase an already high pill burden and result in poor adherence. Moreover, the evidence base to guide depression treatment among hemodialysis patients is limited. In the investigators' previous work, they developed methods to use latent variables and structural equation modeling to isolate depressive symptoms. Other investigators have demonstrated that directly observed treatment enhances the effectiveness of tuberculosis and HIV treatment.

Investigators now propose a cross-sectional study (Phase 1) followed by a single-arm clinical trial (Phase 2) at 17 dialysis facilities. The cross-sectional study will involve assessments of depressive symptoms (using the PHQ-9 screening instrument) as well as dialysis-related complications, anxiety, and quality of life (Quality of Life Questionnaire) in about 1083 patients. Investigators will then use structural equation modeling to develop and validate a hemodialysis-specific PHQ-9 (hdPHQ-9) that will isolate depressive symptoms. The trial will involve 96 patients with confirmed depression who will be assigned to directly observed weekly antidepressant treatment with fluoxetine. The primary outcome of the trial will be remission of depression at 12 weeks. The trial results will also be used to compare the responsiveness of the PHQ-9 and the hdPHQ-9. Investigators anticipate that the hdPHQ-9 will be a valid and responsive instrument that will isolate depressive symptoms in hemodialysis patients and ultimately improve the screening and diagnosis of depression. Investigators also expect that directly observed weekly fluoxetine treatment will be an effective way to manage depression among hemodialysis patients.

DETAILED DESCRIPTION:
Depression is present in about 20-30% of hemodialysis patients and is associated with morbidity and mortality. However, depression is inadequately diagnosed and treated among dialysis patients. This is due in part to the overlap between depressive symptoms (e.g. appetite change, trouble sleeping, feeling tired) and symptoms related to persistent metabolic derangements in hemodialysis patients (e.g. nausea, nocturnal cramps, feeling washed out after treatment). The overlap between depressive symptoms and dialysis complications makes it difficult to diagnose and therefore to treat depression. In addition, prescription of antidepressant medication may increase an already high pill burden and result in poor adherence. Moreover, the evidence base to guide depression treatment among hemodialysis patients is limited. In the investigators' previous work, they developed methods to use latent variables and structural equation modeling to isolate depressive symptoms. Other investigators have demonstrated that directly observed treatment enhances the effectiveness of tuberculosis and HIV treatment.

Investigators now propose a cross-sectional study (Phase 1) followed by a single-arm clinical trial (Phase 2) at 17 dialysis facilities. The cross-sectional study will involve assessments of depressive symptoms (using the PHQ-9 screening instrument) as well as dialysis-related complications, anxiety, and quality of life (Quality of Life Questionnaire) in about 1083 patients. The investigators will then use structural equation modeling to develop and validate a hemodialysis-specific PHQ-9 (hdPHQ-9) that will isolate depressive symptoms. The trial will involve 96 patients with confirmed depression who will be assigned to directly observed weekly antidepressant treatment with fluoxetine. The primary outcome of the trial will be remission of depression at 12 weeks. The trial results will also be used to compare the responsiveness of the PHQ-9 and the hdPHQ-9.

The investigators anticipate that the hdPHQ-9 will be a valid and responsive instrument that will isolate depressive symptoms from dialysis complications and ultimately improve the screening and diagnosis of depression. They also expect that directly observed weekly fluoxetine treatment will be an effective way to manage depression among hemodialysis patients.

Innovative features of the proposed project include the use of latent variables to address overlap, administration of a long acting weekly antidepressant, and directly observed treatment. The project has the potential not only to improve the diagnosis and management of depression among hemodialysis patients but also to improve their morbidity and mortality. Furthermore, it may serve as a model for future studies to isolate symptoms among overlapping medical conditions.

Aim A. To develop and validate a self-reported depression screening instrument that isolates depressive symptoms from hemodialysis-related complications.

Hypothesis: A hemodialysis-specific PHQ-9 (hdPHQ-9) will isolate depressive symptoms from dialysis complications.

Aim B. To determine the impact of directly observed weekly fluoxetine treatment on remission of depression among hemodialysis patients.

Hypothesis: About half of patients who have directly observed fluoxetine treatment will have remission of depression.

Aim C. To examine the responsiveness of the new depression screening instrument to depression treatment.

Hypothesis: Fluoxetine treatment will be associated with larger improvements in hdPHQ-9 scores than in PHQ-9 scores.

ELIGIBILITY:
Inclusion Criteria:

* currently on hemodialysis at a CDC dialysis unit
* English speaking
* able to provide informed consent

Exclusion Criteria:

* on hemodialysis for less than 3 months
* comorbid psychotic, bipolar, substance use dependence, Alzheimer's or dementia

Not eligible for Phase II (intervention) if currently on antidepressant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ash Seghal, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen SD, Norris L, Acquaviva K, Peterson RA, Kimmel PL. Screening, diagnosis, and treatment of depression in patients with end-stage renal disease. Clin J Am Soc Nephrol. 2007 Nov;2(6):1332-42. doi: 10.2215/CJN.03951106. Epub 2007 Oct 17. PMID 17942763
- [Background] Hedayati SS, Bosworth HB, Kuchibhatla M, Kimmel PL, Szczech LA. The predictive value of self-report scales compared with physician diagnosis of depression in hemodialysis patients. Kidney Int. 2006 May;69(9):1662-8. doi: 10.1038/sj.ki.5000308. PMID 16598203
- [Background] Watnick S, Wang PL, Demadura T, Ganzini L. Validation of 2 depression screening tools in dialysis patients. Am J Kidney Dis. 2005 Nov;46(5):919-24. doi: 10.1053/j.ajkd.2005.08.006. PMID 16253733
- [Background] Cohen SD, Kimmel PL. Nutritional status, psychological issues and survival in hemodialysis patients. Contrib Nephrol. 2007;155:1-17. doi: 10.1159/000100952. PMID 17369709
- [Background] Kimmel PL, Peterson RA, Weihs KL, Simmens SJ, Alleyne S, Cruz I, Veis JH. Multiple measurements of depression predict mortality in a longitudinal study of chronic hemodialysis outpatients. Kidney Int. 2000 May;57(5):2093-8. doi: 10.1046/j.1523-1755.2000.00059.x. PMID 10792629
- [Background] Kimmel PL, Peterson RA, Weihs KL, Simmens SJ, Boyle DH, Verme D, Umana WO, Veis JH, Alleyne S, Cruz I. Behavioral compliance with dialysis prescription in hemodialysis patients. J Am Soc Nephrol. 1995 Apr;5(10):1826-34. doi: 10.1681/ASN.V5101826. PMID 7787151
- [Background] Lacson E Jr, Bruce L, Li NC, Mooney A, Maddux FW. Depressive affect and hospitalization risk in incident hemodialysis patients. Clin J Am Soc Nephrol. 2014 Oct 7;9(10):1713-9. doi: 10.2215/CJN.01340214. Epub 2014 Oct 2. PMID 25278546
- [Background] Lopes AA, Albert JM, Young EW, Satayathum S, Pisoni RL, Andreucci VE, Mapes DL, Mason NA, Fukuhara S, Wikstrom B, Saito A, Port FK. Screening for depression in hemodialysis patients: associations with diagnosis, treatment, and outcomes in the DOPPS. Kidney Int. 2004 Nov;66(5):2047-53. doi: 10.1111/j.1523-1755.2004.00977.x. PMID 15496178
- [Background] Chiu YW, Teitelbaum I, Misra M, de Leon EM, Adzize T, Mehrotra R. Pill burden, adherence, hyperphosphatemia, and quality of life in maintenance dialysis patients. Clin J Am Soc Nephrol. 2009 Jun;4(6):1089-96. doi: 10.2215/CJN.00290109. Epub 2009 May 7. PMID 19423571
- [Derived] Kauffman KM, Dolata J, Figueroa M, Gunzler D, Huml A, Pencak J, Sajatovic M, Sehgal AR. Directly Observed Weekly Fluoxetine for Major Depressive Disorder Among Hemodialysis Patients: A Single-Arm Feasibility Trial. Kidney Med. 2022 Jan 17;4(3):100413. doi: 10.1016/j.xkme.2022.100413. eCollection 2022 Mar. PMID 35386606

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screened Via Chart Abstraction 1588 In person Screening Conducted 1248 Evaluated for Major Depression Disorder 110 Untreated for Major Depressive Disorder 27 Consented/enrolled into trial 16
Period: Overall Study
Arm/Group | Fluoxetine Group
Started | 16
Completed | 15
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fluoxetine Group
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
PATIENT HEALTH QUESTIONNAIRE 9 [Mean (Standard Deviation); unit: units on a scale] — 9 questions to gauge depression/depressive symptoms. Each question asks - Over the last 2 weeks, how often have you been bothered by any of the following problems: Each questions 0-3 scale (0=not at all 1= several days 2= more than half the days 3=nearly every day ). Range =0min to 27max.
  A TOTAL SCORE OF ≥10 IS AN ESTABLISHED THRESHOLD FOR CLINICALLY RELEVANT DEPRESSIVE SYMPTOMS.
  units on a scale | 11.3 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Impact of Directly Observed Weekly Fluoxetine Treatment on Remission of Depression Among Hemodialysis Patients.
Description: remission of depression, defined as a week 12 Patient Health Questionnaire 9 (PHQ-9) total score of <5. The survey consists of 9 questions to gauge depression/depressive symptoms. Each question asks - Over the last 2 weeks, how often have you been bothered by any of the following problems: Each questions 0-3 scale (0=not at all 1= several days 2= more than half the days 3=nearly every day ). Range =0min to 27max.
  A TOTAL SCORE OF ≥10 IS AN ESTABLISHED THRESHOLD FOR CLINICALLY RELEVANT DEPRESSIVE SYMPTOMS. Less than 5 is total remission of depressive symptoms.
Time Frame: 3 years
Population: Enrolled 16
  * 13 Female
  * 13 African American
  * 1 Hispanic
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluoxetine Group
Number analyzed (Participants) | 16
units on a scale | 6.6 (2)

ADVERSE EVENTS:
Time Frame: All side effects ASSESSED EVERY OTHER WEEK OVER A TWELVE WEEK PERIOD while patients were actively taking fluoxetine.
Description: Participants will be seen on a weekly basis. Every other week, the study nurse practitioner will review any side effects the participant is having and record any adverse events. These check ins will be recorded on the study Progress Note and also the Fluoxetine Follow Up Checklist form. These notes will be reviewed on a weekly basis by the study team as a whole.
Arm/Group | Fluoxetine Group
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 1/16
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoxetine Group (N=16)
Nausea (Gastrointestinal disorders) | 1 (1) — One individual had stomach pains/nausea after taking the 20 mg fluoxetine and withdrew from the project. This is a common side effect of fluoxetine.

LIMITATIONS AND CAVEATS:
The study sample size is small for multiple reasons, including more patients than anticipated scoring below the threshold on the PHQ-9 or already being on psychiatric medications before enrollment.

conditions. There was no comparison group. As a result, we are unable to compare efficacy and safety with other treatments or to evaluate the potentially confounding effect of frequent interactions with the psychiatric nurse practitioner.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT03390933/Prot_003.pdf
  • Statistical Analysis Plan (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT03390933/SAP_004.pdf
  • Informed Consent Form (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT03390933/ICF_002.pdf